CLINICAL TRIAL: NCT06542731
Title: Phase 1 Study of ONO-4578 Given as Combinations of ONO-4578, ONO-4538, Docetaxel and Ramucirumab in Subjects With Metastatic Non-small Cell Lung Cancer Who Have Had Disease Progression During or After One Prior First-line Anti-PD-(L) 1 Antibody and Platinum-based Chemotherapy for Advanced/Metastatic Disease
Brief Title: An Open-label, Uncontrolled Study of ONO-4578 and ONO-4538 in Combination With Standard-of-care Docetaxel and Ramucirumab as Second-line Therapy in Patients With Advanced or Recurrent Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4578-05
Record Dates: First submitted 2024-08-01; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Docetaxel; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ONO-4578＋ONO-4538＋docetaxel ＋ ramucirumab (Experimental)
  Interventions: Drug: ONO-4578; Drug: ONO-4538; Drug: Docetaxel; Drug: Ramucirumab

INTERVENTIONS:
Drug: ONO-4578 — Specified dose on specified days
Drug: ONO-4538 — Specified dose on specified days
  Other Names: Nivolumab
Drug: Docetaxel — Specified dose on specified days
  Other Names: Taxotere
Drug: Ramucirumab — Specified dose on specified days
  Other Names: Cyramza

SUMMARY:
This study is PhaseⅠstudy to evaluate the tolerability and safety of ONO-4578 and ONO-4538 in combination with standard-of-care docetaxel and ramucirumab as second-line therapy in patients with advanced or recurrent NSCLC who were refractory to a combination therapy containing an anti-PD-(L)1 antibody and a platinum-based drug

ELIGIBILITY:
Inclusion Criteria:

1. Clinical stage III B/ III C with unsuitable for radical irradiation, Clinical stage IV or recurrent non-small cell lung cancer
2. Life expectancy of at least 3 months
3. Patients with ECOG performance status 0 or 1

Exclusion Criteria:

1. Patients with severe complication
2. Patients with multiple primary cancers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-09-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities（DLT） | 21 days
Adverse event(AE) | Up to 28 days after the last dose

SECONDARY OUTCOMES:
Pharmacokinetics（Plasma concentration of ONO-4578） | Up to 28 days after the last dose
Pharmacokinetics（serum concentration of ONO-4538） | Up to 28 days after the last dose
Overall response rate (ORR) | Up to 2 years
Disease control rate (DCR) | Up to 2 years
Overall survival (OS) | Up to 2 years
Progression-free survival (PFS) | Up to 2 years
Duration of response (DOR) | Up to 2 years
Time to response (TTR) | Up to 2 years
Best overall response (BOR) | Up to 2 years
Percentage of change in the sum of tumor diameters of target lesions | Up to 2 years
Maximum percentage of change in the sum of tumor diameters of target lesions | Up to 2 years
Changes in tumor markers（CYFRA,CEA,SLX） | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (13):
- Japan (13):
  - Saitama Cancer Center, Shinden, Saitama
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - Juntendo University Hospital, Bunkyō City
  - Teikyo University Hospital, Itabashi-ku
  - Japan Anti-Tuberculosis Association Fukujuji Hospital, Kiyose-shi
  - The Cancer Institute Hospital of JFCR, Kōtoku
  - Niigata Cancer Center Hospital, Niigata
  - Hyogo Medical University Hospital, Nishinomiya-shi
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute, Osaka
  - Kitasato University Hospital, Sagamihara-shi
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakai
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki-shi
  - Kanagawa Cancer Center, Yokohama

IPD SHARING:
Plan to Share IPD: No